CLINICAL TRIAL: NCT03048279
Title: Registry for Multiple Endocrine Neoplasia Syndromes: MEN1/MEN2
Status: Active, not recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: RCR01-485; NCI-2021-12213 (Other: NCI CTRP Clinical Trials Reporting Registry)
Record Dates: First submitted 2017-02-07; First posted 2017-02-09 (Estimated); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Multiple Endocrine Neoplasia Syndromes
Keywords: Multiple Endocrine Neoplasia Syndromes; MEN1; MEN2; Relatives; Database; Questionnaires; Surveys
MeSH Terms: conditions — Multiple Endocrine Neoplasia | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Multiple Endocrine Neoplasia Syndromes: MEN1/MEN2: Consented individuals will be interviewed by phone and/or mail to obtain medical history specific to their diagnosis of either MEN1 or MEN2.
  Interventions: Behavioral: Questionnaires
- Close Relatives of Registered MDACC MEN Patients: Participants will be asked to complete a health and family history questionnaire. This questionnaire process may be completed by phone or mail.
  Interventions: Behavioral: Questionnaires

INTERVENTIONS:
Behavioral: Questionnaires — Multiple Endocrine Neoplasia Syndromes: MEN1/MEN2 Group: Participants interviewed by phone and/or mail to obtain medical history specific to their diagnosis of either MEN1 or MEN2.
  Close Relatives of Registered MDACC MEN Patients Group: Participants asked to complete a health and family history questionnaire. This questionnaire process may be completed by phone or mail.
  Other Names: Surveys

SUMMARY:
Objectives:

To contribute new and prospective data to our existing database library for patients with MEN1 and MEN2 at The University of Texas M.D. Anderson Cancer Center.

DETAILED DESCRIPTION:
Previously followed MEN1 and MEN2 patients at M.D. Anderson Cancer Center will be mailed an introductory letter and a "consent to be contacted" form to determine whether they are interested in participating in the study. New MEN1 and MEN2 patients seen in clinic at M.D. Anderson Cancer Center will be asked if they wish to learn more about this study. Interested patients will also be asked to distribute the introductory letter and consent to be contacted form to their blood relatives. Printed materials regarding this study will only be mailed to non-MDACC individuals with the expressed written or verbal permission from a consenting MDACC patient. All interested individuals will return the signed "consent to be contacted" form to the PI. Consented individuals will be interviewed by phone and/or mail to obtain updated family and medical history specific to their diagnosis of either MEN1 or MEN2. To verify accuracy of medical data collected, all non-MDACC participants will be asked if they consent to have their off-site medical records released to us for review. There will be no treatment or collection of blood or tissue in this study.

Although this study presents minimal risk to participants, participant consent will be obtained due to the need to obtain permission to make contact with patients and their families.

Approximately 1500 patients and their relatives will be included in this study. This will be done on an inpatient and outpatient basis.

ELIGIBILITY:
Inclusion Criteria:

1. Registered MDACC patients diagnosed with MEN1 or MEN2.
2. Close relatives of registered MDACC MEN patients.

Exclusion Criteria:

1. Individuals who are either non-MDACC registered patients or do not have a close relative who is an MEN patient registered at MDACC.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: MEN1 and MEN2 patients at M.D. Anderson Cancer Center and their relatives
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2001-09-05 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Contribution of New and Prospective Data to Existing Database Library for Patients with MEN1 and MEN2 by Completion of Health Questionnaires | 25 years

CONTACTS AND LOCATIONS:
Overall Officials: Nancy D. Perrier, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center — http://www.mdanderson.org